CLINICAL TRIAL: NCT04068883
Title: Controlled DTI Evaluations in High School Football and Female Soccer to Evaluate Efficacy of Jugular Compression Collar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-1123
Record Dates: First submitted 2018-12-27; First posted 2019-08-28 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: MTBI - Mild Traumatic Brain Injury; Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collar group (Experimental): group of athletes that will wear the collar device
  Interventions: Other: Q collar
- Non Collar group (No Intervention): group of athletes that will not wear the collar device

INTERVENTIONS:
Other: Q collar — An externally-worn medical device that applies mild jugular compression
  Arms: Collar group

SUMMARY:
The purpose of the study is to monitor longitudinal changes in brain structure between the preseason and postseason, in a population of football and soccer playing athletes wearing the Device and compared to a similar population not wearing the device. Secondly, the purpose is to determine the efficacy of device to reduce alterations in brain structure relative to amount and magnitude of sustained head impacts. Finally, to show that DTI efficacy and safety results can be prospectively confirmed in a multi-school investigation.

Test the null hypotheses of no difference between collar users and non-collar users changes from baseline to end of season for:

* Primary: Alterations in pre-defined DTI metrics (AD, MD, RD) are significantly reduced in the neck collar group at EOS relative to BL.
* Secondary: Alterations in pre-defined DTI metrics is explained by the number of hits, the hit intensity, and the intensity per head impact over the season non-collar users.

In addition, secondary analytics on data derived from injury surveillance (musculoskeletal, concussion and symptom/severity scores), behavioral (Trail Making, Postural Sway, Flanker, Task-switching, Near Point Convergence, ADHD and King Devick) or imaging (DTI, fMRI, T1, T2, and MRS) will be evaluated.

DETAILED DESCRIPTION:
Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). A simple, effective, and lightweight device worn by athletes or war fighters in the field, designed to mitigate TBI resulting from blast trauma or concussive events, would save lives, and the huge costs incurred for life-treatment of surviving victims. An externally-worn medical device that applies mild jugular compression according to the principle of the Queckenstedt Maneuver (the Device) is being developed by Q30 Sports Science, LLC (Q30). Preliminary research indicates that the Device has the potential to reduce the likelihood of alterations to brain microstructure. The currently developed collar has been approved for studies in humans and the results indicate safety for use during high demand and maximal exertion activities, Study IDs: 2013-2240, 2016-7948, 2014-5009, 2016-9625, 2016-0988, and 2015-2205 Institutional Review Board - Federalwide Assurance #00002988). FDA has determined that this device is a nonsignificant risk (NSR) device study because it does not meet the definition of a significant risk (SR) device under § 812.3(m) of the investigational device exemptions (IDE) regulation (21 CFR 812).

This study will investigate the effectiveness of this device in high school athletes playing a collision sport such as football or soccer. Athletes participating in this study will be randomly assigned to one of two groups: 1) Device wearing during the season or 2) Non-device wearing during the season. Male football players and female soccer players will be included in this investigation. All participants may be outfitted with an accelerometer which will measure the magnitude of every impact to the head sustained by the athlete. This accelerometer will be affixed with an adhesive patch,(which will be placed behind the ear, to measure the magnitude of every impact to the head sustained by the athlete Effectiveness of the device will be determined via differences in longitudinal brain imaging and behavioral assessments following competitive football and soccer participation. The investigators will also enroll a group of athletes involved in a non-contact sport (such as cross-country) to act as controls.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Able to provide written consent
* Must be 13 years or older and a participant on a high school football or soccer team

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or severe head trauma as indicated through pre-season screening:
* Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Any known airway obstruction
* Any known seizure disorder
* Prothrombotic or hyperthrombotic condition
* Cerebral cavernous malformation
* Players not medically cleared to play sports

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 488 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
TBSS measured change in axial diffusivity pre to post season | 6 months
  Alterations in pre-defined DTI metrics (AD, MD, RD) are significantly reduced in the neck collar group at EOS relative to BL.
TBSS measured change in radial diffusivity pre to post season | 6 months
  Alterations in pre-defined DTI metrics (AD, MD, RD) are significantly reduced in the neck collar group at EOS relative to BL.
TBSS measured change in mean diffusivity pre to post season | 6 months
  Alterations in pre-defined DTI metrics (AD, MD, RD) are significantly reduced in the neck collar group at EOS relative to BL.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinnati Childrens Hospital
Locations (2):
- United States (2):
  - Cincinanti Childrens Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT04068883/ICF_001.pdf
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT04068883/Prot_002.pdf